CLINICAL TRIAL: NCT01514409
Title: Sub-chronic Effects of 5-hydroxytryptophan on Mood and Emotional Processing in Healthy Volunteers: A Randomised Trial
Brief Title: Sub-chronic Effects of 5-hydroxytryptophan on Mood and Emotional Processing in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24AQ1
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Mood
Keywords: 5-hydroxytryptophan; Mood; Emotional Processing; Emotional Cognition; Nutritional Supplement; Low mood
MeSH Terms: conditions — Consciousness Disorders | interventions — 5-Hydroxytryptophan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-Hydroxytryptophan (Experimental)
  Interventions: Dietary Supplement: 5-Hydroxytryptophan
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Pharmaceutical grade silica

INTERVENTIONS:
Dietary Supplement: 5-Hydroxytryptophan — Thirty-three participants were randomly allocated in a double-blind manner to receive either 3x50mg capsules of 5-HTP or placebo (silica) for 14 days.
  5-HTP is produced commercially by extraction from the seeds of the African plant griffonia simplicifolia.
  Arms: 5-Hydroxytryptophan
Dietary Supplement: Pharmaceutical grade silica — Pharmaceutical grade silica was utilized as placebo
  Arms: Placebo

SUMMARY:
5-hydroxytryptophan (5-HTP) is a nutritional supplement sold in many health food stores, and is taken in order to raise levels of serotonin in the brain. Serotonin is a neurotransmitter that is involved in the regulation of mood.

Previous research has assessed the effects of raising serotonin levels using tryptophan (the precursor of 5-HTP) and serotonergic antidepressants on emotional processing in healthy volunteers. However, to date there has been no human trial investigating the effects of 5-HTP on emotional processing in healthy volunteers.

Thus, the current study aims to assess the effects of 5-HTP, on emotional processing and mood in healthy volunteers.

DETAILED DESCRIPTION:
The serotonin precursor 5-HTP is sold as a nutritional supplement and has been used to offset low mood for over 30 years due to its ability to raise levels of neural serotonin. However, evidence for the efficiency of 5-HTP is limited and the mechanism of action of 5-HTP in offsetting low mood has not been well-characterised.

The current study assessed the ability of 5-HTP to induce biases for positive emotional material in healthy volunteers, similar to those induced by serotonergic antidepressants and the nutritional supplement tryptophan. The effects of 5-HTP on subjective mood and depressive symptoms were also assessed.

Participants were randomised to receive either 150mg of 5-HTP or placebo daily for 14 days. Depressive symptoms and subjective mood were assessed pre- and post-intervention. Emotional processing was assessed on the 15th day using a battery of emotionally valenced cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* Healthy
* Aged 18-65
* Not taking any herbal or prescription medications (excluding contraceptive pill)
* Free from depressive illness or mood disorder for the last 6 months
* Free of physical illness

Exclusion Criteria:

* Physically ill
* History of medical illness
* Current or previous (6 month) history of psychiatric disorder
* Pregnant/breastfeeding
* Allergy or hypersensitivity to any of the ingredients contained in the investigational product
* Taking any medication (excluding contraceptive pill)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | 14 days
  The BDI-II is a measure used to assess the severity of depressive symptoms. It is comprised of 21 items that are scored on a scale ranging from 0-3, with total scores ranging from 0-63. Scores of over 16 are indicative of depressive symptoms.
Profile of Mood States-Bipolar (POMS-BI) | 14 days
  The POMS-BI is a measure used to assess subjective mood. It comprises 72 adjectives which describe mood states. Participants indicate how well the adjectives describe how they feel on a four point scale ranging from 0-3. The POMS-BI measures the following six bipolar mood states: composed-anxious, elated-depressed, agreeable-hostile, clearheaded-confused, energetic-tired, and confident-unsure.
Emotional Perception: Facial Expression Recognition Task | 14 days
  Participants are shown faces displaying five different emotions - happiness, sadness, fear, anger, and disgust. Each facial expression has been morphed between 0% (neutral) to 100% in 25% increments. Four examples of each emotion at each intensity are displayed on a computer screen (84 stimuli presentations in total). Faces are displayed for 500ms aand then replaced with a blank screen. Participants have to indicate what facial expression has been displayed by clicking the corresponding button on-screen with the mouse. Accuracy, reaction times, and misclassifications are measured.
Emotional Categorisation and Memory | 14 days
  Participants are shown sixty personality characteristics consecutively (30 agreeable, 30 disagreeable)on a computer screen in random order for 500ms each. Participants are asked to judge whether the personality traits are 'likeable' or 'dislikeable'. Classifications and reaction times for correct choices are recorded. Participants are then asked to recall as many personality characteristics as they can in order to assess their incidental memory for positive versus negative material.
Emotional Attention: Attentional Probe Task | 14 days
  The attentional probe task based on MacLeod, Matthews and Tata's (1986) visual attention paradigm is used to assess participants attention towards positive versus negatively valenced words. Accuracy and reaction time is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom